CLINICAL TRIAL: NCT04656470
Title: Neuroimaging Study of Dexmedetomidine-Induced Analgesia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Oluwaseun Johnson-Akeju, MD, MMSc, Associate Professor of Anaesthesia, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2019P000996
Record Dates: First submitted 2020-10-01; First posted 2020-12-07 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-10

CONDITIONS: Analgesia; Anesthesia
MeSH Terms: conditions — Agnosia | interventions — Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: Patients will receive dexmedetomidine anesthesia during the study visit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dexmedetomidine (Experimental): During the study visit, patients will be delivered dexmedetomidine anesthesia. 0.5mcg/kg of dexmedetomidine solution will be infused over 10 minutes, and then up to 0.5mcg/kg/hr will be maintained for an additional 20-30 minutes.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Patients will be delivered dexmedetomidine anesthesia to gain greater understanding of its analgesic effects.
  Other Names: Precedex

SUMMARY:
Neuroimaging data will be collected for patients that are given low doses of dexmedetomidine in order to understand its analgesic effects.

DETAILED DESCRIPTION:
In this trial, participants will be given dexmedetomidine using a single-arm study design. fMRI will be conducted during this time. Cognitive assessments and pain monitoring will be administered at various points before and after dexmedetomidine is administered.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 to 45
* Normal body weight and habitus, BMI ≤ 30
* Non-smoker
* American Society of Anesthesiologists (ASA) physical status classification P1
* Active health insurance coverage
* Fully vaccinated against COVID-19

Exclusion Criteria:

* Cardiovascular: myocardial infarction, coronary artery disease, peripheral vascular disease, arrhythmia, congestive heart failure, valvular disease, hypertension
* Respiratory: bronchitis, chronic obstructive pulmonary disease, smoking, shortness of breath
* Hepatic: hepatitis, jaundice, ascites
* Neurologic: seizure, stroke, positive neurologic findings on neurologic examination, multiple sclerosis, Meniere's disease, Parkinson's disease, neuropathy, peripheral stenosis
* Gastrointestinal: esophageal reflux, hiatal hernia, ulcer
* Endocrine: diabetes, thyroid disease
* Renal: acute or chronic severe renal insufficiency
* Hematologic: blood dyscrasias, anemia, coagulopathies, on anticoagulant therapy
* Musculoskeletal: prior surgery or trauma to head neck or face, arthritis, personal or family history of malignant hyperthermia
* Psychiatric: history or treatment for an active psychiatric problem, depression
* Reproductive: pregnancy, breast-feeding
* Medications: regular use of prescription and non-prescription medications expected to affect CNS function, St. John's Wort
* Allergies: dexmedetomidine, ondansetron, glycopyrrolate, phenylephrine
* Dermatologic: ulcerative skin conditions or other dermatologic conditions which could interfere with blood pressure cuff placement.
* MRI reasons for exclusion: History of head trauma, surgical aneurysm clips, cardiac pacemaker, prosthetic heart valve, neurostimulator, implanted pumps, cochlear implants, metal rods, plates, or screws, intrauterine device, hearing aid, dentures, metal injury to eyes, metallic tattoos anywhere on the body or near the eye.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2022-03-04 (Actual); Primary Completion 2025-05-27 (Actual); Study Completion 2025-05-27 (Actual)

PRIMARY OUTCOMES:
Effect of Dexmedetomidine on Pain Processing Circuitry | Change in brain functional connectivity between baseline pain and dexmedetomidine pain during the fMRI visit, an average of 90 minutes
  fMRI data will be used to compare changes in brain connectivity due to pain using functional network and seed-based correlation analyses when a pain cuff (Hokanson Rapid Cuff Inflator) is inflated during baseline and dexmedetomidine analgesia periods.

CONTACTS AND LOCATIONS:
Overall Officials: Oluwaseun Johnson-Akeju, MD, MMSc, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No